CLINICAL TRIAL: NCT00883246
Title: Determination of Effectiveness of SilverHawk Peripheral Plaque Excision (SilverHawk Device) for the Treatment of Infrainguinal Vessels/Lower Extremities
Brief Title: Study of SilverHawk®/TurboHawk® in Lower Extremity Vessels (DEFINITIVE™ LE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Endovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEFINITIVE LE
Record Dates: First submitted 2009-04-16; First posted 2009-04-17 (Estimated); Results first posted 2015-10-09 (Estimated); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Peripheral Arterial Disease; Claudication; Critical Limb Ischemia
Keywords: PAD
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Chronic Limb-Threatening Ischemia | interventions — Atherectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Atherectomy (Other): All patients enrolled in this single-arm study were treated with directional atherectomy.
  Interventions: Device: SilverHawk & TurboHawk Peripheral Plaque Excision System

INTERVENTIONS:
Device: SilverHawk & TurboHawk Peripheral Plaque Excision System — Removal of atherosclerotic plaque from artery walls.
  Other Names: SilverHawk (Atherectomy), TurboHawk (Atherectomy)

SUMMARY:
The purpose of the study is to evaluate the intermediate and long-term effectiveness of stand-alone atherectomy treatment of peripheral arterial disease in the legs.

ELIGIBILITY:
Inclusion Criteria

* Has a Rutherford Clinical Category Score of 1 - 6.
* Has evidence of ≥ 50% stenosis or occlusion in the superficial femoral, popliteal, anterior tibial, posterior tibial and/or peroneal arteries, confirmed by angiography.
* Has identifiable distal target vessel which upon completion of the intervention, is anticipated to provide re-constitution of blood flow to the foot.
* Exchangeable guidewire must cross lesion(s), with ability of catheter to cross lesion.
* Each discrete target lesion's length is ≤ 20 cm.
* Reference vessel diameter is ≥ 1.5 mm and ≤ 7 mm.

Exclusion Criteria

* Has surgical or endovascular procedure of the target vessel within 14 days prior to the index procedure.
* Has any planned surgical intervention or endovascular procedure within 30 days after the index procedure.
* Has had a previous peripheral bypass affecting the target limb.
* Has end-stage renal disease defined as undergoing hemodialysis for kidney failure.
* Has presence of severe calcification in target lesion(s).
* Has in-stent restenosis of the target lesion.
* Has an aneurysmal target vessel.
* Has significant stenosis or occlusion of inflow tract that has not been revascularized prior to treatment of the target vessel.
* Has perforation, dissection or other injury of the access or target vessel requiring additional stenting or surgical intervention prior to enrollment.
* Has disease that precludes safe advancement of the SilverHawk/TurboHawk device to the target lesion(s).
* Has had a previous amputation above the metatarsal line on the target limb.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2009-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Garcia, MD, Principal Investigator — St. Elizabeth's Medical Center, Tuft's University School of Medicine; James McKinsey, MD, Principal Investigator — The New York Presbyterian/Columbia University; Professor Thomas Zeller, Principal Investigator — Herz-Zentrum Bad Krozingen Germany

REFERENCES:
- [Background] McKinsey JF, Zeller T, Rocha-Singh KJ, Jaff MR, Garcia LA; DEFINITIVE LE Investigators. Lower extremity revascularization using directional atherectomy: 12-month prospective results of the DEFINITIVE LE study. JACC Cardiovasc Interv. 2014 Aug;7(8):923-33. doi: 10.1016/j.jcin.2014.05.006. PMID 25147039

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with all severities of peripheral arterial disease were recruited for this single-arm study. Outcome measures may apply to all subjects or be specific to level of disease severity (ie subjects w/claudication RCC1-3, subjects w/critical limb ischemia RCC4 (no wounds) or RCC5-6 (with wounds)). These are specified in the Arm/Group titles.
Pre-assignment Details: 800 subjects were enrolled. One subject was excluded from all data analyses due to an invalid informed consent and was not considered started.
Groups:
- Atherectomy: All patients enrolled in this single-arm study were treated with directional atherectomy.
  SilverHawk Peripheral Plaque Excision System: Removal of atherosclerotic plaque from artery walls.
Period: Overall Study
Arm/Group | Atherectomy
Started | 799
Completed | 626
Not Completed | 173

BASELINE CHARACTERISTICS:
Population: 800 patients were enrolled, but 1 subject's data were excluded from all analyses due to an invalid informed consent, yielding a cohort of 799 analyzable subjects.
Arm/Group | Atherectomy
Number analyzed (Participants) | 799
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 259
  >=65 years | 540
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.1 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 363
  Male | 436
Region of Enrollment [Number; unit: participants]
  Europe | 107
  United States | 692
Diabetes [Number; unit: participants]
  Diabetes | 418
  No Diabetes | 381

OUTCOME MEASURES:

1. Primary Outcome: Primary Patency Rate (in Patients Treated for Claudication RCC 1-3)
Description: The primary endpoint analysis for claudication subjects was primary patency rate at one year, defined by duplex ultrasound measurement of peak systolic velocity ratio ≤ 3.5 at the target lesion(s) with no clinically-driven reintervention within the treated segment in subjects who had claudication (RCC of 1 - 3) at time of enrollment.
Time Frame: One year
Population: Kaplan-Meier estimate of the freedom from loss of primary patency in lesions (N=743 lesions)
Measure: Number; unit: percentage of lesions by Kaplan Meier
Units Other Than Participants: Number of Lesions Analyzed
Groups:
- Claudicant Subgroup: Subjects who had claudication (RCC of 1 - 3) at time of enrollment.
Arm/Group | Claudicant Subgroup
Number analyzed (Participants) | 598
Number analyzed (Number of Lesions Analyzed) | 743
percentage of lesions by Kaplan Meier | 81.6

2. Primary Outcome: Amputation-Free Survival at 1 Year (in Patients Treated for Critical Limb Ischemia RCC 4-6)
Description: The primary endpoint for CLI was amputation-free survival at one year, defined as freedom from a major, unplanned amputation of the target limb through the 1-year visit in subjects who have CLI (RCC 4 - 6) at time of enrollment.
Time Frame: One Year
Measure: Number; unit: percentage of subjects by Kaplan-Meier
Groups:
- CLI Subgroup: Subjects who had CLI (RCC 4 - 6) at time of enrollment
Arm/Group | CLI Subgroup
Number analyzed (Participants) | 201
percentage of subjects by Kaplan-Meier | 95.1

3. Secondary Outcome: Device Success (in All Patients Enrolled)
Description: Device success was defined as ≤ 30% residual stenosis following use of the SilverHawk device, as measured by angiography, without adjunctive endovascular interventions or periprocedural complications.
Time Frame: Immediately following use of the SilverHawk device
Population: Lesions with core angiographic laboratory measurements of residual stenosis
Measure: Number; unit: percentage of Lesions
Units Other Than Participants: Number of Lesions Analyzed
Groups:
- All Patients: All patients enrolled in this single-arm study were treated with directional atherectomy.
  SilverHawk Peripheral Plaque Excision System: Removal of atherosclerotic plaque from artery walls.
Arm/Group | All Patients
Number analyzed (Participants) | 799
Number analyzed (Number of Lesions Analyzed) | 999
percentage of Lesions | 70.5

4. Secondary Outcome: Procedural Success (in All Patients Enrolled)
Description: Procedure success was defined as ≤ 30% residual stenosis following use of SilverHawk device and adjunctive endovascular interventions (if required) as measured by angiography without periprocedural complications.
Time Frame: Immediately following use of the SilverHawk and adjunctive devices
Population: All lesions with angiographic core lab assessment of residual stenosis at the end of the procedure were included
Measure: Number; unit: percentage of lesions
Units Other Than Participants: Number of Lesions Analyzed
Arm/Group | All Patients
Number analyzed (Participants) | 799
Number analyzed (Number of Lesions Analyzed) | 1015
percentage of lesions | 84.0

5. Secondary Outcome: Major Adverse Event Rate (in All Patients Enrolled)
Description: Major Adverse Event Rate (MAE) at 30 Days was defined as clinically-driven target vessel revascularization (TVR), major unplanned amputation of treated limb, or all-cause mortality within 30 days post procedure, as classified by the Clinical Events Committee (CEC).
Time Frame: 30 Days
Measure: Number; unit: percentage of patients
Arm/Group | All Patients
Number analyzed (Participants) | 799
percentage of patients | 1.6

6. Secondary Outcome: Major Adverse Event Rate (in All Patients Enrolled)
Description: Major Adverse Event Rate at One Year was defined as clinically-driven target vessel revascularization, major unplanned amputation of the treated limb, or all-cause mortality within one year, as classified by the Clinical Events Committee (CEC).
Time Frame: One Year
Measure: Number; unit: percentage of patients
Arm/Group | All Patients
Number analyzed (Participants) | 799
percentage of patients | 20.9

7. Secondary Outcome: Improvement in Walking Impairment Questionnaire Score (in Patients Treated for Claudication RCC 1-3)
Description: WIQ includes a measurement for walking distance, walking speed, and climbing stairs collected at baseline and one year, presented for subjects who have claudication. The Walking Improvement Questionnaire (WIQ) is a validated method to assess objective improvement in functional walking ability of subjects with intermittent claudication. Difficulty walking a distance was self-assessed at baseline by the patient (prior to treatment) and at the one year follow up visit. Speed and stair climbing ability were assessed by the treating physician. Scale ranges from 0 (minimum) to 100 (maximum), with larger numbers representing better outcomes. An increase in WIQ scores at 1 year represents an improvement over baseline.
Time Frame: Baseline and 1 Year
Population: All subjects treated for claudication RCC 1-3 with completed WIQ forms
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Claudicant Subgroup (Baseline): All claudicant subjects enrolled in this single-arm study were treated with directional atherectomy and had walking distance measured prior to treatment.
  SilverHawk Peripheral Plaque Excision System: Removal of atherosclerotic plaque from artery walls.
- Claudicant Subgroup (One Year): All claudicant subjects (RCC 1-3) enrolled in this single-arm study were treated with directional atherectomy and walking distance measured at the one year follow-up visit.
  SilverHawk Peripheral Plaque Excision System: Removal of atherosclerotic plaque from artery walls.
Arm/Group | Claudicant Subgroup (Baseline) | Claudicant Subgroup (One Year)
Number analyzed (Participants) | 590 | 464
units on a scale
  Walking Distance Score | 19.9 (24.2) | 49.5 (38.0)
  Walking Speed Score: number analyzed (Participants) | 582 | 441
  Walking Speed Score | 20.3 (20.7) | 39.4 (28.8)
  Stair Climbins Score: number analyzed (Participants) | 574 | 448
  Stair Climbins Score | 32.0 (31.0) | 53.9 (37.6)

8. Secondary Outcome: Improvement in Rutherford Clinical Category (in All Patients Enrolled)
Description: Change in RCC at One Year was assessed and percentage of subjects with an improvement in clinical status indicated by a decrease of one or more in RCC at one year compared to baseline, that is attributable to the treated limb (in cases of bilateral disease), was calculated.
Time Frame: 1 Year
Population: All patients with RCC data at baseline and 1 year
Measure: Number; unit: percentage of patients
Arm/Group | All Patients
Number analyzed (Participants) | 616
percentage of patients | 82.3

9. Secondary Outcome: Ankle-Brachial Index (in All Patients Enrolled)
Description: Change in Ankle-Brachial Index at One Year was calculated and percentage of subjects with an increase (improvement) in the ankle-brachial index (ABI) at one year compared to baseline in subjects with compressible arteries and baseline ABI < 0.9 was calculated.
Time Frame: 1 Year
Population: All patients with compressible arteries and a baseline ABI < 0.9.
Measure: Number; unit: percentage of patients improved
Arm/Group | All Patients
Number analyzed (Participants) | 429
percentage of patients improved | 76

10. Secondary Outcome: Secondary Patency (in Patients Treated for Claudication RCC 1-3)
Description: Secondary patency was defined as measured by duplex ultrasound peak systolic velocity ratio ≤ 3.5 maintained by repeat percutaneous intervention in subjects who have claudication; estimated as freedom from loss of patency by the Kaplan-Meier method at one year.
Time Frame: One Year
Population: All claudicants.
Measure: Number; unit: percentage of lesions
Units Other Than Participants: Number of Lesions Analyzed
Arm/Group | Claudicant Subgroup
Number analyzed (Participants) | 598
Number analyzed (Number of Lesions Analyzed) | 743
percentage of lesions | 93.5

11. Secondary Outcome: Primary Patency (in Patients Treated for Critical Limb Ischemia RCC 4-6)
Description: The primary patency for CLI was defined by duplex ultrasound measurement of peak systolic velocity ratio ≤ 3.5 at the target lesion(s) with no clinically-driven reintervention within the treated segment in subjects who have CLI at time of enrollment
Time Frame: One Year
Population: All patients with CLI.
Measure: Number; unit: percentage of lesions
Units Other Than Participants: Number of Lesions Analyzed
Arm/Group | CLI Subgroup
Number analyzed (Participants) | 201
Number analyzed (Number of Lesions Analyzed) | 279
percentage of lesions | 74.1

12. Secondary Outcome: Amputation-Free Survival (in Patients Treated for Claudication RCC 1-3)
Description: Amputation-Free Survival in Claudicants at One Year was defined as freedom from a major, unplanned amputation of the target limb through the one year visit in subjects who have claudication at time of enrollment.
Time Frame: One Year
Population: All claudicants.
Measure: Number; unit: percentage of patients by Kaplan-Meier
Groups:
- Claudicant Subjects: Subjects who had claudication (RCC of 1 - 3) at time of enrollment.
Arm/Group | Claudicant Subjects
Number analyzed (Participants) | 598
percentage of patients by Kaplan-Meier | 99.6

13. Secondary Outcome: Improvement in Wound Healing (in Patients Treated for Critical Limb Ischemia and With Wounds RCC 5-6)
Description: Wound healing at three months was defined as a decrease of at least one Wagner Classification grade of the wound at three months compared to baseline in subjects who have Rutherford Clinical Category score of 5 or 6 at the time of enrollment.
Time Frame: 3 months
Population: Patients with wounds at baseline who had wound assessment scores at baseline and at 3 months.
Measure: Number; unit: percentage of patients
Groups:
- CLI Subgroup: Wound healing was assessed in subjects who had Rutherford Clinical Category score of 5 or 6 at the time of enrollment.
Arm/Group | CLI Subgroup
Number analyzed (Participants) | 103
percentage of patients | 61.2

14. Secondary Outcome: Alternative Patency Rate (Peak Systolic Velocity ≤ 2.4) at 1 Year (in Patients Treated for Claudication RCC 1-3)
Description: Defined by the duplex ultrasound measurement of peak systolic velocity ration ≤ 2.4 at the target lesion (s) with no clinically-driven re- intervention with the treated segment in subjects who have claudication at time of enrollment.
Time Frame: 1 year
Population: Lesions in patients with claudication at baseline
Measure: Number; unit: percentage of lesions by Kaplan-Meier
Units Other Than Participants: Number of Lesions Analyzed
Arm/Group | Claudicant Subgroup
Number analyzed (Participants) | 598
Number analyzed (Number of Lesions Analyzed) | 743
percentage of lesions by Kaplan-Meier | 77.5

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the 12 month follow-up of the study.
Description: Adverse events were reviewed and classified by a third party clinical events committee. AEs were classified as device-related and/or procedure-related, as well as Serious Adverse Events (SAEs) and Major Adverse Events (MAEs).
Arm/Group | All Patients
All-Cause Mortality (participants affected / at risk) | 4/799
Serious Adverse Events (participants affected / at risk) | 410/799
Other Adverse Events (participants affected / at risk) | 41/799
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=799)
Abrupt closure (Vascular disorders) | 3 (4)
Access site complication (Vascular disorders) | 16 (16)
Arterial dissection (Grade D or greater) (Vascular disorders) | 5 (5)
Arterial Spasm (Vascular disorders) | 3 (3)
Arterial thrombosis (Vascular disorders) | 9 (10)
Arterio-venous fistula (Vascular disorders) | 1 (1)
Bleeding complications (Vascular disorders) | 11 (12)
Cellulitis (Vascular disorders) | 5 (5)
Hypertension (Vascular disorders) | 1 (1)
Hypotention (Vascular disorders) | 4 (4)
Infection (not at access site) (Infections and infestations) | 48 (70)
Myocardial Infarction (Vascular disorders) | 17 (18)
Other (Vascular disorders) | 279 (458) — Other" included events such as acute coronary syndrome, back pain, fractures, cancers, non-target lesions revascularizations, heart failure, pneumonia, etc.
Pseudoaneurysm not at the access site (Vascular disorders) | 1 (1)
renal failure (Renal and urinary disorders) | 8 (8)
Renal Insufficiency (Renal and urinary disorders) | 1 (1)
Restenosis (Vascular disorders) | 170 (218)
Sepsis (Infections and infestations) | 7 (9)
stroke (Vascular disorders) | 7 (7)
Sub-acute Closure (Vascular disorders) | 1 (1)
Tansient ischemic attack (Vascular disorders) | 6 (6)
Wound abscess (Infections and infestations) | 1 (1)
wound debridement (Surgical and medical procedures) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=799)
Arterial perforation (Vascular disorders) | 41 (42)

LIMITATIONS AND CAVEATS:
The study's principal limitations include a lack of randomization and follow-up beyond 12 months.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less